CLINICAL TRIAL: NCT06118814
Title: Investigation of Virtual Reality Supported Core Stabilization Exercises and Basic Body Awareness Therapy Activities in Individuals With Adolescent Idiopathic Scoliosis
Brief Title: Body Awareness in Adolescent Idiopatic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Ertugrul Deniz Kose, Phd Student, Hitit University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HititUni
Record Dates: First submitted 2023-10-29; First posted 2023-11-07 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Scoliosis Idiopathic Adolescent; Body Image
Keywords: Scoliosis Idiopathic Adolescent; Body Awareness; Virtual Reality Exercise
MeSH Terms: interventions — Exergaming

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Body Awareness Therapy Group (Experimental): In addition to the home program, basic body awareness exercises will be applied.
  Interventions: Other: Body Awareness Therapy Exercise; Other: Home Exercise
- Virtual Reality Exercise Group (Experimental): In addition to the home program, virtual reality-supported core stabilization exercises will be applied.
  Interventions: Other: Virtual Reality Exercise; Other: Home Exercise
- Core Stability Exercise Group (Experimental): In addition to the home program, core stabilization exercises will be performed.
  Interventions: Other: Core Stability Exercise; Other: Home Exercise
- Home Exercise Group (Active Comparator): A home program will be implemented.
  Interventions: Other: Home Exercise

INTERVENTIONS:
Other: Body Awareness Therapy Exercise — Body awareness therapy exercises were applied to the subjects in this group.
  Arms: Body Awareness Therapy Group
Other: Virtual Reality Exercise — Virtual reality exercises were applied to the subjects in this group.
  Arms: Virtual Reality Exercise Group
Other: Core Stability Exercise — Core stabilization exercises were applied to the subjects in this group.
  Arms: Core Stability Exercise Group
Other: Home Exercise — Subjects in this group implemented a home exercise program.

SUMMARY:
Scoliosis is a three-dimensional deformity of the spine, and Adolescent Idiopathic Scoliosis (AIS) is the most common subtype of scoliosis. There are various scoliosis-specific exercise programs available for the treatment of scoliosis, and core stabilization is one of the methods aimed at maintaining spinal alignment.

Virtual reality offers a method to create stimulating and engaging environments using task-oriented techniques to increase individual interest and motivation. In the literature, virtual reality applications have been used in healthcare to facilitate recovery, post-morbid rehabilitation, and to improve performance in athletes. However, there is limited research on the application of virtual reality therapy for scoliosis patients. One study mentioned the use of two scoliosis-specific exercises through video-assisted games, but the limited exercise repertoire did not make a significant difference. Other video-assisted studies have suggested that exercises targeting posture, balance, and gait can be used for scoliosis patients. Therefore, our study aims to apply core stabilization exercises to scoliosis patients using virtual reality applications and investigate their effects on patient development.

Although studies examining the effectiveness of core stabilization exercises on body awareness in adolescents with idiopathic scoliosis are limited, they have been reported to be effective in terms of pain, body image, quality of life and functionality.

This study aims to benefit from the therapeutic effects and contribute to the literature by using both different treatment methods. There are four groups in the study. Each group will be evaluated before and after ten weeks of treatment. Participants diagnosed with adolescent idiopathic scoliosis will be randomly assigned to three groups for the study. All participants will be evaluated before and after treatment for curvature severity and rotation angle, trunk flexibility, trunk normal joint range of motion, spine pain, Cosmetic Defect Assessment-Walter Reed Visual Assessment Scale (WRVAS), Quality of Life Assessment-"Scoliosis Research Association-22" (SRS-22) and Child Depression Scale (CDI).

DETAILED DESCRIPTION:
After the power analysis, it was planned to include 40 individuals in our study, 10 individuals in each group. The groups of this study will be as follows:

* First group, virtual reality-supported core stabilization exercises (stability-enhancing exercises for the muscles around the spine) and additional home program group,
* Second group, core stabilization exercises (stability-enhancing exercises for the muscles around the spine) and additional home program group,
* Third group, basic body awareness treatment techniques and additional home program group,
* Fourth group is only home program treatment group. The treatment program is planned as a total of 20 sessions for 10 weeks, two days a week. This study was planned as single-blind to ensure the impartiality of the evaluation.

All individuals and their parents who will participate in the study will be verbally informed about the content of the study, its duration, the evaluations to be made, the treatments to be applied and the expected goals to be achieved. Signed consent forms will be obtained from the individuals and their parents indicating that they are willing to participate in the study. The sociodemographic information, physical characteristics, short leg length, age at scoliosis diagnosis, Cobb angle at first diagnosis, curve type and location results of all individuals participating in the study will be recorded. Individuals who do not want to continue the study will be excluded from the study. The study will be completed and the results will be evaluated after the final evaluations of the individuals continuing the study are completed. All participants will be re-evaluated before and after the treatment for their curve severity and rotation angle, trunk flexibility, trunk normal joint range of motion, spinal pain, the Walter Reed Visual Assessment Scale (WRVAS), the Quality of Life Assessment Scale (SRS-22), and the Children's Depression Scale (CDI).

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 10 and 18, having a diagnosis of AIS (Adolescent Idiopathic Scoliosis),
* not using a brace,
* having a Cobb angle between 10º-40º,
* being able to regularly attend the prescribed program,
* not having any pulmonary or thoracic cage-related diseases such as rib fractures, atelectasis, or asthma, not having any neurological or psychiatric disorders, and not having a chronic condition requiring medication, and obtaining parental consent for the child's participation in the program.

Exclusion Criteria:

* The patient should not have any contraindications for exercise,
* should not have received any scoliosis treatment or undergone spinal surgery within the last year,
* should not be using a brace,
* should not have scoliosis limited only to the cervical region,
* should not have any neuromuscular, cardiovascular, or respiratory function disorder, and should not have cognitive impairment.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-08-10 (Actual)

PRIMARY OUTCOMES:
Cobb Angle | Up to 3 months
  Measurements are made to grade scoliosis using the frontal plane radiography using the Cobb method.

SECONDARY OUTCOMES:
Walter Reed Visual Assessment Scale | Up to 3 months
  It is a scale developed to evaluate the physical deformity perceived by patients with scoliosis.
Scoliosis Research Society Questionnare | Change from pre treatment and post treatment.
  It is a simple and practical quality of life questionnaire created specifically for individuals with scoliosis. It includes parameters of pain, self-image/appearance, function/activity, mental health, and treatment satisfaction.
Spinal Pain Assessment | Up to 3 months
  Visual Analog Scale will be used to evaluate spinal pain.
Trunk Muscle Endurance Assessment | Up to 3 months
  Straight plank and side plank tests will be used to evaluate trunk muscle endurance.
Trunk Muscle Strength Assessment | Up to 3 months
  "sit-up test" and "modified push-up test" will be used to evaluate trunk flexor and extensor muscle strength.
Balance Assessment | Up to 3 months
  Y balance balance test will be used for dynamic balance measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- Hitit University, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No